CLINICAL TRIAL: NCT06663540
Title: Synergies Between Physical Exercise and the Abacus and Their Effects on Improving Academic Learning and Well-being in Childhood.
Brief Title: Synergies Between Exercise and Abacus in Childhood.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University A
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Childhood
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group that will continue with their usual school routine
- Experimental Group (Experimental): The experimental group will participate in weekly sessions that integrate physical exercise and the use of the abacus. This will include physical activities such as sports, outdoor games or physical education classes, for approximately two hours a week. In addition, they will receive teaching sessions that incorporate the abacus to develop mathematical and problem-solving skills.
  Interventions: Other: Exercise & Abacus

INTERVENTIONS:
Other: Exercise & Abacus — Features two main interventions: physical exercise sessions and abacus training activities.
  Physical Exercise Sessions aim to enhance fitness and cognitive function through activities like aerobic exercises and team sports. Research indicates that regular physical activity can improve memory, attention, and problem-solving skills essential for academic success.
  Abacus Training Activities focus on developing mathematical skills and cognitive abilities. Children learn to manipulate the abacus for calculations, which enhances numerical understanding and memory retention, positively impacting academic performance.
  The program's innovative dual approach suggests that integrating physical and cognitive training can lead to greater improvements in academic performance and emotional resilience than either intervention alone.
  Arms: Experimental Group

SUMMARY:
This study investigates the synergistic effects of physical exercise and abacus training on enhancing academic performance and well-being in children. It aims to establish a comprehensive educational framework that leverages the cognitive benefits of both physical activity and mental math skills. Research indicates that regular physical exercise not only contributes to better physical health but also significantly enhances cognitive functions such as memory, attention, and problem-solving abilities. Studies have shown that active children tend to perform better academically due to improved brain function and increased focus. Simultaneously, abacus training has been recognized for its role in developing mathematical skills and cognitive abilities. It promotes visual-spatial reasoning and enhances memory retention, which can lead to better performance in mathematics and related subjects.

By integrating these two methods, seeks to provide children with a holistic approach to learning, fostering not only academic success but also emotional and psychological resilience. Preliminary findings suggest that children engaged in combined physical and cognitive training programs show notable improvements in their academic outcomes and overall well-being compared to those who participate in traditional learning environments. The project emphasizes the importance of creating educational strategies that prioritize comprehensive child development, suggesting that a balanced approach involving both physical exercise and cognitive training tools like the abacus can lead to significant benefits in children's learning experiences.

ELIGIBILITY:
Inclusion Criteria:

* School-aged children, ages 6-7.
* Students who are able to engage in moderate-intensity physical activity without medical restrictions and are able to handle the abacus.
* Students who can regularly participate in the intervention program sessions and follow-up assessments.
* Voluntary participation, with informed consent signed by parents or legal guardians.

Exclusion Criteria:

* Children with health conditions that prevent them from safely engaging in physical activity or using the abacus (e.g., heart disease, severe respiratory problems, motor disabilities that limit physical activity).
* Students with severe cognitive or learning disabilities that may significantly interfere with the use of the abacus or the ability to equitably benefit from the intervention.
* Children who are unable to commit to continued participation in the program, whether for personal or logistical reasons.
* Students who are involved in other extracurricular or school programs focused on cognitive or physical training, to avoid overlapping effects of other interventions.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Self-Concept | Up to twelve weeks
  The perception children have of themselves, influencing their motivation and learning strategies. Measured using the Self-Concept Scale for Children, scores range from 20 to 80, with scores below 50 indicating low self-concept, scores between 50-70 indicating average self-concept, and scores above 70 indicating a high self-concept.
Self-Esteem | Up to twelve weeks
  Refers to the value and respect children have for themselves. The Rosenberg Self-Esteem Scale will be utilized, where scores range from 0 to 30. A score below 15 indicates low self-esteem, scores between 15-25 suggest moderate self-esteem, and scores above 25 indicate high self-esteem.
Attention | Up to twelve weeks
  The ability to focus on specific stimuli while ignoring distractions. Attention levels will be assessed using the Test of Variables of Attention, with a scoring range of 0 to 100. A score below 70 suggests attention deficits, while scores between 70-85 indicate average attention, and scores above 85 suggest above-average attention.
Concentration | Up to twelve weeks
  The capacity to maintain focus over extended periods. The Concentration Test measures children's ability to concentrate, with scores ranging from 0 to 100. Scores below 60 indicate poor concentration, 60-80 suggest average concentration, and scores above 80 indicate strong concentration abilities.
Creativity | Up to twelve weeks
  The ability to think outside the box and generate new ideas. The Torrance Tests of Creative Thinking will be employed, where scores range from 0 to 100. Scores below 60 indicate low creativity, 60-80 suggest average creativity, and scores above 80 indicate high creativity.
Physical Well-Being | Up to twelve weeks
  Encompasses overall physical health, including fitness levels. Measured using the Physical Fitness Test, which provides a composite score from various fitness activities. A score below the 50th percentile indicates below-average physical fitness, while scores above the 50th percentile indicate average or above-average physical fitness.
Mental Well-Being | Up to twelve weeks
  Refers to emotional health and the ability to cope with stress. The General Health Questionnaire will be utilized, where scores range from 0 to 36. A score above 12 suggests potential mental health issues, scores between 6-12 indicate moderate mental well-being, and scores below 6 indicate good mental health.
Cognitive Performance | Up to twelve weeks
  Involves skills such as memory and problem-solving, assessed using the Wechsler Intelligence Scale for Children. The total IQ score ranges from 40 to 160, where scores below 70 indicate intellectual disability, scores between 70-85 indicate borderline intellectual functioning, and scores above 85 indicate average or above-average cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No